CLINICAL TRIAL: NCT07331519
Title: Integrating Smoking Cessation With Low-dose CT-screening for Lung Cancer - a Randomized Study
Brief Title: Integrating Smoking Cessation With Low-dose CT-screening for Lung Cancer
Acronym: ISC-LDCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Collaborators: Finnish Cancer Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EETMK 15/2025; EETMK 15/2025 (Other: Ethics Committee of the Wellbeing Services County of North Ostrobothnia)
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-02

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; lung cancer; low-dose CT; lung cancer screening
MeSH Terms: conditions — Smoking Cessation; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Smoking cessation with a smartphone application + LDCT lung cancer screening
  Interventions: Other: Smartphone application; Other: low-dose computed tomography
- Arm 2 (Active Comparator): Smoking cessation with written materials + LDCT lung cancer screening
  Interventions: Other: low-dose computed tomography; Other: Written materials for smoking cessation
- Arm 3 (Active Comparator): Smoking cessation with a smartphone application without LDCT lung cancer screening
  Interventions: Other: Smartphone application

INTERVENTIONS:
Other: Smartphone application — Suunta smartphone application for smoking cessation
  Arms: Arm 1; Arm 3
Other: low-dose computed tomography — Low-dose computed tomography based screening for lung cancer
  Arms: Arm 1; Arm 2
Other: Written materials for smoking cessation — Written materials for smoking cessation
  Arms: Arm 2

SUMMARY:
The study investigates effectiveness of different smoking cessation methods and low-dose CT based lung cancer screening

DETAILED DESCRIPTION:
The study population consists of individuals aged 50-74 years with a significant smoking history who continue to smoke. The study design is a prospective and participants are randomized into three study arms: low-dose CT (LDCT) + smoking cessation with a smartphone application (arm 1), LDCT + smoking cessation with written materials (arm 2), smoking cessation with a smartphone application without LDCT (arm 3). The study compares effectiveness of smoking cessation methods, LDCT in lung cancer screening, lung cancer stage distribution, and lung cancer specific survival.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent
2. Age between 50-74
3. Smoked ≥ 15 cigarettes/day for ≥ 25 years or smoked ≥ 10 cigarettes/day for ≥ 30 years and are active smokers (smoking during the last two weeks)
4. Access to a smartphone (iPhone or Android)

Exclusion Criteria:

1. Current or past melanoma, lung, renal or breast cancer
2. A chest CT examination less than one year before inclusion
3. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
4. No access to a smartphone (iPhone or Android)
5. Participant is unwilling or unable to comply with treatment and trial instructions
6. Any condition that study investigators consider an impediment to safe trial participation

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2036-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of smoking cessation | three months
  The percentage of participants who have quitted smoking between the study arms 1 vs. 2

SECONDARY OUTCOMES:
Rate of smoking cessation | Three months
  The percentage of participants who have quitted smoking between all the study arms
Rate of smoking cessation | 12 and 24 months
  The percentage of participants who have quitted smoking between all the study arms
Rate of long-term smoking cessation | 12 and 24 moths
  The percentage of participants who have had abstinence of smoking for at least six months
LDCT findings | baseline and 24 months
  The percentage of LDCT negative, indetermined, and positive findings by screening round
Sensitivity and specificity of LDCT screening examination | 24 months, 36 months, and 10 years
  Sensitivity and specificity of LDCT screening examination for lung cancer detection (arms 1&2 vs. 3)
Lung cancer incidence | 24 months, 36 months, and 10 years
  Lung cancer incidence (stage specific) (arms 1&2 vs. 3)
Frequency of self-reported smoking cessation verified with CO measurement | 24 months
  Frequency of self-reported smoking cessation verified with CO measurement

CONTACTS AND LOCATIONS:
Overall Officials: Tytti Särkeälä, PhD, Study Director — Finnish Cancer Society
Locations (5):
- Finland (5):
  - Helsinki University Hospital, Helsinki
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
  - Vaasa Central Hospital, Vaasa

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in this article will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available beginning 6 months after publication and ending 3 years thereafter.
Access Criteria: Data will be shared with qualified researchers who submit a methodologically sound proposal for analyses that align with the original study aims. Proposals should be submitted to the corresponding author. Access will require a data use agreement.

REFERENCES:
- [Result] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Result] de Koning HJ, van der Aalst CM, de Jong PA, Scholten ET, Nackaerts K, Heuvelmans MA, Lammers JJ, Weenink C, Yousaf-Khan U, Horeweg N, van 't Westeinde S, Prokop M, Mali WP, Mohamed Hoesein FAA, van Ooijen PMA, Aerts JGJV, den Bakker MA, Thunnissen E, Verschakelen J, Vliegenthart R, Walter JE, Ten Haaf K, Groen HJM, Oudkerk M. Reduced Lung-Cancer Mortality with Volume CT Screening in a Randomized Trial. N Engl J Med. 2020 Feb 6;382(6):503-513. doi: 10.1056/NEJMoa1911793. Epub 2020 Jan 29. PMID 31995683
- [Result] Iivanainen S, Kurtti A, Wichmann V, Andersen H, Jekunen A, Kaarteenaho R, Vasankari T, Koivunen JP. Smartphone application versus written material for smoking reduction and cessation in individuals undergoing low-dose computed tomography (LDCT) screening for lung cancer: a phase II open-label randomised controlled trial. Lancet Reg Health Eur. 2024 May 25;42:100946. doi: 10.1016/j.lanepe.2024.100946. eCollection 2024 Jul. PMID 39070744